CLINICAL TRIAL: NCT00246467
Title: A Phase 1b, Multi-Centre, Parallel Group, Single Blind Study to Evaluate the Safety, Tolerability and Immunogenicity of a Recombinant Plague Vaccine (rF1 and rV Antigens) in Healthy Subjects
Brief Title: One Year Study to Evaluate Three Different Adjuvanted Doses of the Recombinant Plague Vaccine (rF1 and rV Antigens)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAthene UK Limited (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05-0005; AVEC/rYP/03
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Plague
Keywords: plague
MeSH Terms: conditions — Plague | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Alhydrogel
Biological: rF1 and rV protein antigens

SUMMARY:
One hundred and five subjects will be recruited into three groups. Each subject will receive two doses of recombinant plague vaccine at one of three dose levels (rF1 and rV recombinant antigen proteins).

DETAILED DESCRIPTION:
Plague is an infection occurring in small rodents and mammals caused by the gram-negative bacterium Yersinia pestis (Y. pestis). Transmission from rodent to man is usually by a flea vector leading to the characteristic swelling of the lymph nodes draining the region of the bite, followed by a septicaemic illness (classic bubonic plague). Human-to-human transmission can occur via droplet nuclei spread by coughing of patients with bubonic or septicaemic plague who have developed pulmonary lesions (pneumonic plague). However, cases of pulmonary transmission have also been described from household pets. In pneumonic plague symptoms of a respiratory infection develop first followed by an acute onset septicaemic illness. In the military context, the likely exposure is via the inhalation route, as a Biological Warfare Agent (BWA), and therefore protection against pneumonic plague is the paramount requirement. This is a phase 1, parallel group, single-blind study of 105 healthy adult aged 18-55, randomly assigned to one of the three cohorts and will receive the same dose of vaccines (2x) and then re-randomized at 6 months to receive either a third dose or placebo, in order to determine the safety and tolerability associated with different primary immunization doses of recombinant IM plague vaccine (rF1 and rV) antigen proteins for optimum safe dose, assess responses (both antibody and cell-mediated) following immunization, investigate the correlation between cell-mediated and antibody titers and to assess the duration of the immune responses to antigens following a third dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females.
2. Aged between 18-55 years (inclusive) on Day 0 of the Study.
3. Of a body mass index (BMI) of 18-35 inclusive.
4. Able to understand the informed consent form and other documents required to be read by the subject.
5. Willing to give signed informed consent
6. Able to give a medical history without major organ pathology (e.g. cardiac, immunological, psychiatric, endocrine or neurological disorders, cancer or other wasting diseases - (adequately treated actinic keratosis, or basal cell carcinoma [BCC], or carcinoma in situ [CIS] of the cervix are permitted).
7. In the case of female subjects, they may be enrolled if one of the following criteria applies:

   Either Is not pregnant or breast feeding AND is routinely using adequate injectable or transdermal (administered at the recommended frequency) or oral contraception (at a stable dose for at least three months prior to the first dose of vaccine) and will continue to do so during the study, augmenting this contraceptive measure with a barrier method OR is sexually abstinent OR is monogamous and has a partner who has had a vasectomy (>1 month previously) OR is using a commonly recognised copper and hormone implanted intrauterine device (IUD) such as TCu-380A, TCu-220C, MLCu-375, Nova-T or LNG-20. In addition, the subject must have a negative blood pregnancy test prior to enrolment into the study (see also Criterion 9 below).

   Or Is post menopausal (defined as a female with no menstrual cycle for at least the previous 24 months AND is of menopausal age (>45 years) Or Has not had a menstrual cycle for between 12 and 24 months AND is of menopausal age (>45 years) AND has had a negative blood pregnancy test prior to enrolment into the study and a negative urine pregnancy test pre-dose.

   Or Has been surgically sterilised (confirmed by review of medical record). Or Has had a total hysterectomy at least 3 months prior to the start of the study (confirmed by review of medical record).
8. A male may be enrolled if willing to use barrier methods of contraception and whose partner is using an acceptable form of contraception for 3 months after each dose.
9. A female subject must have a negative urine pregnancy test prior to each dosing (unless post-menopausal, surgically sterilised, or has had a total hysterectomy, as defined in Criterion 7 above).
10. 12-lead electrocardiogram (ECG) recording without signs of pathology and conduction disturbances and with a QTc interval of < 450 msec for males and < 470 msec for females. ECGs will be analysed automatically for study entry purposes and will also be analysed by a cardiologist within 24 hours. QT intervals will be recorded automatically by the ECG machines used.

Exclusion Criteria:

1. Presence of any clinically significant medical condition as determined by the Investigator.
2. History of clinically significant hypersensitivity or idiosyncratic reaction related to any medical product, including vaccines and aminoglycoside antibiotics (such as kanamycin).
3. History or evidence of drug misuse.
4. Participation in a clinical study of an investigational vaccine within 3 months prior to the start of the study (Day 0) or an investigational drug product within 30 days prior to the start of the study.
5. Use of any prescription or non-prescription medication within 7 days prior to the first dosing with the exception of over-the-counter (OTC) antihistamines, non-steroidal anti-inflammatory drugs (NSAID) including aspirin, acetaminophen, OTC decongestants, herbal medicines (except St. John's Wort), oral/injectable/transdermal contraceptives, OTC multi-vitamin preparations (not high-dose preparations) or oral iron supplements. Any medication taken within 7 days of the first dosing will be documented.
6. History or suspicion of inability to co-operate adequately.
7. Donation of blood or blood products during the 4 weeks prior to participation in the study (Day 0).
8. Immunodeficiency or clinically active autoimmune disease.
9. Positive urine alcohol and/or drug screen for drugs of misuse (opiates, methadone, cocaine, amphetamines, cannabinoids, and barbiturates).
10. Positive serological test for human immunodeficiency virus (HIV), and/or hepatitis B virus and/or hepatitis C virus.
11. Vaccination(s) with a live vaccine in the 4 weeks prior to participation in the study, (or 'flu vaccine in the 2 weeks prior to participation), or killed / inactivated / sub-unit vaccines in the previous 3 weeks.
12. Receipt of blood or plasma transfusions, or pooled gamma globulin, in the 3 months prior to participation in the study (Day 0) and/or a need for future blood or plasma transfusions during this study.
13. Prior receipt of any plague vaccine.
14. Prior history of plague infection (confirmed or suspected) or significant exposure to Y. pestis (e.g. a laboratory worker who regularly handles Y. pestis) as judged by the investigator.
15. Clinically relevant abnormal findings on routine physical examination.
16. Clinically significant out-of-range laboratory tests at screening including: urinalysis, serum creatinine, serum electrolytes (sodium, potassium, chloride and bicarbonate), liver function tests (ALT, AST and GGT), lactate dehydrogenase (LDH), white blood cell count, absolute neutrophil count, platelet count, clotting and blood haemoglobin. Minor, out-of-range laboratory test results for the above tests may be allowable, at the discretion of the Investigator, if such results are within 10% of the normal ranges and considered to be not clinically significant.
17. Twelve-lead ECG recording with clinically relevant signs of pathology and conduction disturbances as judged by the investigator.
18. Presence of tattoos that cover or partially cover the upper arm, and which would limit adequate assessment of the injection site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2005-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety of recombinant plague vaccine

SECONDARY OUTCOMES:
Immunogenicity of recombinant plague vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Clinical Research
Locations (10):
- United States (9):
  - Accelovance, Huntsville, Alabama
  - Accelovance, Washington D.C., District of Columbia
  - Florida Medical Research Institute, Gainesville, Florida
  - Accelovance, Melbourne, Florida
  - Miami Research Associates, Miami, Florida
  - Radiant Research, Pinellas Park, Florida
  - Accelovance, South Bend, Indiana
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Accelovance, Amarillo, Texas
- Simbec Research Limited, Merthyr Tydfil, United Kingdom